CLINICAL TRIAL: NCT00465660
Title: The Effect of 6 Month High Intensity Progressive Resistance Training on Knee Articular Cartilage Morphology in Female Osteoarthritic Patients
Brief Title: Resistive Exercise for Arthritic Cartilage Health (REACH)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACTRN012605000116628
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2006-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Cartilage; Exercise; Progressive Resistance Training
MeSH Terms: conditions — Osteoarthritis; Motor Activity

INTERVENTIONS:
Behavioral: Progressive resistance training

SUMMARY:
Female subjects over the age of 40 will be recruited and randomised into a progressive resistance training (PRT) or sham-exercise group. The PRT group will train at 80% of their peak strength, using Keiser pneumatic resistance machines, and progress approximately 3% per session. Strength will be re-assessed fortnightly. Exercises will target muscles around the hip and knee. The sham-exercise group will train on the same equipment as the PRT group except hip adduction, but without added resistance or progression. Both groups will train 3 days per week for roughly 45 minutes for 6 months.

It is hypothesised that high intensity PRT will decelerate the tibial and femoral cartilage degeneration in the knee affected most by OA.

Primary Outcome:

Articular cartilage morphology following 6 months high intensity progressive resistance training

Secondary Outcomes:

Muscle and fat cross-sectional area (CSA) (pre and post) Muscle strength, power, endurance, and contraction velocity (pre, 3 months, & post) Medications (pre, 3 months, & post) Body composition (pre, 3 months, & post) Balance; Physical function (pre, 3 months, & post) Questionnaires (pre, 3 months, & post)

* Habitual exercise (PASE) -WOMAC index (pain, stiffness and functional ability)
* Depressive symptoms (Depression Scale) -Quality of life (SF36)
* Confidence performing physical activity (Ewart) -Demographics

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged over 40 years old
* Primary Osteoarthritis in at least one knee using standard criteria of the American College of Rheumatology (ACR) criteria for classification of clinical osteoarthritis
* Ambulatory without human assistance
* Willingness to be randomised to experiential or control group
* Ability to attend scheduled exercise and testing sessions

Exclusion Criteria:

* Regular exercise of any kind over the past 3 months (>1dpw).
* Secondary osteoarthritis (traumatic or post-surgical), rheumatic disease, gouty or septic arthritis, Paget's disease, pseudogout, major congenital abnormalities, hemochromatosis, Wilson's disease and other rare forms of arthritis
* Joint injury, injection or surgery within the past 6 months or knee joint replacement
* Contraindications to MRI/Exercise

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2009-07

PRIMARY OUTCOMES:
Articular cartilage morphology following 6 months high intensity progressive resistance training

SECONDARY OUTCOMES:
Muscle and fat cross-sectional area (CSA) (pre and post)
Muscle strength, power, endurance, and contraction velocity (pre, 3 months, & post)
Medications (pre, 3 months, & post)
Body composition (pre, 3 months, & post)
Balance; Physical function (pre, 3 months, & post)
Questionnaires (pre, 3 months, & post):
Habitual exercise (PASE)
WOMAC index (pain, stiffness and functional ability)
Depressive symptoms (Depression Scale)
Quality of life (SF36)
Confidence performing physical activity (Ewart)
Demographics

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte Vanwanseele, PhD, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia